CLINICAL TRIAL: NCT02305212
Title: Applying Cogmed to Improve Working Memory Abilities After Traumatic Brain Injury
Brief Title: Cogmed for Working Memory After TBI
Acronym: Cogmed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director, Kessler Foundation
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 786-13 Cog
Record Dates: First submitted 2013-12-19; First posted 2014-12-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Traumatic Brain Injury
Keywords: Working Memory
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cogmed (Experimental): Cogmed is a cognitive rehabilitation protocol designed to improve working memory. The Cogmed sessions are on a computer at home for 30-40 min per day, 5 days per week for 5 weeks.
  Interventions: Behavioral: Cogmed
- Wait list (No Intervention)

INTERVENTIONS:
Behavioral: Cogmed
  Arms: Cogmed

SUMMARY:
This study will examine a cognitive rehabilitation protocol targeted at working memory deficits for adults and children with Traumatic Brain Injury (TBI). In this randomized clinical trial, the efficacy of Cogmed, a cognitive rehabilitation protocol designed to improve working memory, will be examined in children with TBI. Neuropsychological and daily life functioning will be measured. Participants will be children (N=20) and adults (N=20) with a documented history of TBI. Participants will be randomized to a treatment group or a wait list control group. The Experimental Group will receive the Cogmed working memory training program 30-40 minutes per day, 5 days a week for 5 weeks for a total training time of approximately 15 hours. The Control Group will be a wait list control group that will cross over into treatment after the follow-up assessment. All subjects will undergo repeat assessments following completion of the working memory training protocol after the 7th week and again at 13 weeks to document changes in working memory performance.

ELIGIBILITY:
Inclusion Criteria:

* History of Traumatic Brain Injury

Exclusion Criteria:

* Diagnosis of other neurological conditions

Ages: 9 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2016-06-02 (Actual); Study Completion 2016-06-02 (Actual)

PRIMARY OUTCOMES:
Change in scores on standardized tests of working memory | Three points in time: Baseline assessment, Week 7 and Week 13
  Measured via standardized neuropsychological tests (i.e. paper and pencil testing)

SECONDARY OUTCOMES:
Change in scores on self report measures of emotional functioning, assessed via questionnaire | Three points in time: Baseline assessment, Week 7 and Week 13
Change in scores on self report measures of memory functioning, assessed via questionniare | Three points in time: Baseline assessment, Week 7 and Week 13
Change in scores on self report measures of quality of life, assessed via questionnaire | Three points in time: Baseline assessment, Week 7 and Week 13

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Chiaravalloti, Ph.D., Principal Investigator — Kessler Fondation
Locations (2):
- United States (2):
  - Childrens Specialized Hosptial, Mountainside, New Jersey
  - Kessler Foundation, West Orange, New Jersey